CLINICAL TRIAL: NCT06432244
Title: The Effect of the Number of Central Lymph Nodes on Changes in Parathyroid Function
Status: Completed | Type: Observational
Sponsor: Shandong Provincial Hospital (Other Government)
Collaborators: Shandong University (Other)
Responsible Party: Principal Investigator, Guojun Wu, principle investigator, Shandong Provincial Hospital
Other Study IDs: NO.SWYX2024-279
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; central lymph nodes; PTH
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Number of central lymph node dissection: By exploring the relationship between the number of lymph nodes in the central region of the thyroid gland and parathyroid function, evaluate the effectiveness of different surgical procedures and intraoperative protective measures on parathyroid function protection.

SUMMARY:
This study collected data from patients who underwent thyroidectomy in the Breast and Thyroid Surgery Department of Shandong Provincial Hospital from January 2020 to December 2023 by reviewing medical records. The main calculation indicator was the changes in PTH before and after surgery. This study grouped patients based on the number of central lymph nodes under postoperative paraffin pathology, and statistically analyzed the changes and differences in PTH before and after surgery in different groups to verify the relationship between the number of central lymph nodes in the thyroid gland and parathyroid function, and to provide reference for surgical selection in thyroid cancer patients with multiple cervical lymph node metastases.

DETAILED DESCRIPTION:
The central lymph nodes of the thyroid gland refer to the lymph nodes located around the thyroid and trachea. The central lymph nodes are the primary site of thyroid cancer metastasis, and therefore play an important role in thyroid surgery. In thyroid surgery, preventive central lymph node dissection is a routine procedure, but during this process, the parathyroid gland may be impaired due to surgical injury or insufficient blood supply.

Hypothyroidism, also known as parathyroidism, is a common complication of thyroid surgery. When the parathyroid gland is accidentally injured or its blood supply is disrupted, it can lead to insufficient production of parathyroid hormone. Parathyroid hormone is a key hormone that regulates blood calcium levels. Insufficient levels can lead to hypocalcemia, manifested as hand and foot spasms, muscle spasms, and even arrhythmia.

From a surgical perspective, the number of lymph nodes in the central region of the thyroid gland may affect the preservation and functional protection of the parathyroid gland. A large number of lymph nodes indicates that they may have a wider range of disease invasion, requiring more thorough lymph node dissection, thereby increasing the risk of damaging the parathyroid gland or its blood supply.

ELIGIBILITY:
Inclusion Criteria:

* All cases were the first to undergo thyroidectomy surgery.
* All clinical data and research materials of the cases are complete.
* All cases underwent thyroid function examination before and after surgery.
* All cases underwent preoperative thyroid and neck lymph node examinations by the Ultrasound Department of Shandong Provincial Hospital.

Exclusion Criteria:

* Except for cases of recurrence.
* Cases with incomplete clinical data and research materials are excluded.
* Cases that have not undergone thyroid function tests before and after surgery are excluded.
* Excluding cases of secondary surgery.
* Cases that have not undergone thyroid and neck lymph node examinations by the Ultrasound Department of Shandong Provincial Hospital before surgery are excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study collected data from patients who underwent thyroidectomy surgery at the Breast and Thyroid Surgery Department of Shandong Provincial Hospital from January 2020 to December 2023. All patients included in the study had complete clinical data and research materials, with approximately 2000 participants.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
PTH level | 4 weeks
  This study grouped the central lymph nodes based on postoperative paraffin pathology, and statistically analyzed the changes and differences in PTH before and after surgery in different groups to verify the relationship between the number of central lymph nodes in the thyroid gland and parathyroid function.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong provincial hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
The IPD are not publicly available due to privacy and ethical restrictions.